CLINICAL TRIAL: NCT01835730
Title: Phase 1 Multicenter, Randomized, Double-Blind, Placebo Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Response of PE0139 Injection in Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: Phase 1 Multicenter, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Response of PE0139 Injection in Adult Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PE0139-PT-CL-0001
Record Dates: First submitted 2013-03-28; First posted 2013-04-19 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PE0139 Injection (Experimental): Single subcutaneous injection of PE0139, 40 mg/mL
  Interventions: Drug: PE0139 Injection
- Placebo (Placebo Comparator): Single subcutaneous injection of 0.9% Sodium Chloride (NaCl) (Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PE0139 Injection
  Arms: PE0139 Injection
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is a first-in-human randomized, double-blind (Investigator and subject), placebo controlled single ascending dose study that will enroll approximately 40 (6 active/2 placebo per dose group) adult male and female subjects with Type 2 Diabetes Mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent and follow all study-related procedures;
* Male and female subjects at least 18 years of age;
* Male subjects and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their dose of study drug;
* Body mass index ≤45 kg/m2;
* Diagnosed with T2DM and who is currently taking a stable daily dose of a basal insulin (Lantus) plus at least one oral antihyperglycemic agent at a stable dose for 3 months prior to screening.

Exclusion Criteria:

* Currently taking or have taken within 3 months prior to screening an approved or investigational GLP-1 analogue/agonist (e.g., Victoza®) or pramlintide;
* Currently taking or have routinely taken, within 3 months prior to screening , a short-acting insulin;
* Currently taking or have taken, within 3 months prior to screening, a long acting insulin other than Lantus®;
* Known allergy to, or serious adverse effect caused by an approved, or investigational insulin product or any of its components;
* Currently taking any of the following medications: thiazide or furosemide diuretics, beta-blockers, estrogens or other hormonal replacement therapy, or other chronic medications with known adverse effects on glucose tolerance levels unless the subject has been on stable doses of such agents for at least 2 months prior to screening and have no planned changes during the study period;
* History of recurrent severe hypoglycemia (more than 2 episodes within the last 6 months prior to randomization or hypoglycemic unawareness;
* Malignant disease defined as 1) any history of malignant melanoma or breast cancer and/or 2) history of other types of cancer within the last 5 years prior to screening;
* Unstable cardiovascular disease defined as one or more of the following: History of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to screening; History of or currently have New York Heart Association Class III-IV heart failure prior to screening; Uncontrolled/sustained hypertension; History or evidence of long QT syndrome or mean triplicate 12-lead electrocardiogram demonstrating QT interval;
* Clinically significant renal and/or hepatic dysfunction;
* Absolute requirement for corticosteroids or have received systemic steroids within 3 months prior to Randomization (V5, Day -1). Note: Use of inhaled or topical corticosteroids will be permitted;
* Pregnant or lactating female subjects;
* Known history of or active alcohol abuse or use of illicit drugs within 1 year prior to screening;
* Positive screening for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies at V1;
* Participating in any other study and have received any other investigational medication or device within 30 days prior to Visit 1.
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Vital Signs from baseline (Day 0 Pre-dose) | Vital signs Day 0, 1, 2, 3, 4, 5, 6, 7, 14 and 28
  Safety will be evaluated by analyses of the change from baseline in vital signs.
Change in ECGs from baseline (Day -1) | ECG Days 2 and 28
  Safety will be evaluated by analyses of the change from baseline in 12-lead ECG.
Change in Safety Labs from baseline (Pre-dose) | Safety Labs Days 0, 7 and 28
  Safety will be evaluated by analyses of the safety laboratory parameters.
Incidence and severity of immunogenicity | Immunogenicity Days 0, 7, 14 and 28
  Safety will be evaluated by the incidence and severity of immunogenicity.
Incidence and severity of adverse events including hypoglycemia | As reported between Days -10 to 28
  Safety will be evaluated by the incidence and severity of adverse events including hypoglycemia.

SECONDARY OUTCOMES:
Pharmacokinetic Profile | Day 0, 1, 2, 3, 4, 5, 6, and 7
  Pharmacokinetic parameters include: Area under the concentration curve from time 0 to infinity (AUC(0-inf)), Area under the concentration curve to the final sample with a concentration greater than or equal to Limit of Quantitation (LOQ) (AUC(0-t)), Time to maximum concentration (Tmax), Maximum serum concentration (Cmax), Elimination rate constant (Lambda-z), Elimination half-life (t1/2), Clearance uncorrected for bioavailability (CL/F), Distribution uncorrected for bioavailability (Vz/F)
Pharmacodynamic Response | FPG Day -10, -4, 0, 1, 2, 3, 4, 5, 6, 7, and 28; 4-pt Glucose and CGM - Day -10 to -7, -6, -5, and -4 to 7
  To assess the pharmacodynamic response (time action profile) of various single doses of PE0139. Assessments include Fasting plasma glucose (FPG), 4-point serial glucose monitoring and glucose assessed by continuous glucose monitoring (CGM).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brazg, MD, Principal Investigator — Rainier Clinical Research
Locations (3):
- United States (3):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Palm Springs Research Institute, Hialeah, Florida
  - Rainier Clinical Research, Renton, Washington